CLINICAL TRIAL: NCT03918330
Title: Spatial Analysis of the Intestinal Microbiota in Healthy Subjects
Status: Completed | Type: Observational
Sponsor: Örebro University, Sweden (Other)
Collaborators: Region Örebro County (Other)
Responsible Party: Sponsor
Other Study IDs: SpIM
Record Dates: First submitted 2019-04-12; First posted 2019-04-17 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bacterial DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Research on the human intestinal microbiota is common as there is rising evidence of its influence on host physiology and several diseases. Predominantly, it has been based on analyses of faecal samples because of their easy sampling. A minority of studies investigated the gut microbiota using mucosal samples. Not much is known about the spatial differences in microbiota composition along the large bowel. The spatial differences of the gut microbiota without preparation of the bowel have not been analysed yet. Furthermore, the composition of the microbiota of the luminal gut content has not been analysed yet.

This study aims to gain knowledge of the microbial composition of luminal and mucosal samples at different segments of the lower gastrointestinal tract: ileum, caecum, ascending colon, transverse colon, descending colon, sigmoid colon and rectum, as well as of rectal swabs and faecal samples.

DETAILED DESCRIPTION:
The investigators aim to evaluate complete colonoscopies from 10 healthy subjects. This study is used as a first explorative study of how the human gut microbiota is distributed along the lower gastrointestinal tract. No comparable studies in an uncleansed bowel have been performed so far. The number of subjects is based on other studies investigating the microbial composition of mucosal- and faecal-associated microbiota in which a sample size of 10 was enough to detect a difference. An equal number of men and women will be recruited. Drop-outs will be replaced.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Age: 18-65 years

Exclusion Criteria:

1. Known organic gastrointestinal disease (e.g. inflammatory bowel disease, irritable bowel syndrome, chronic diarrhoea or constipation)
2. History of or present gastrointestinal malignancy or polyposis
3. Recent (gastrointestinal) infection (within last 6 months)
4. History of major gastrointestinal surgery (e.g. gastric bypass)
5. Eosinophilic disorders of the gastrointestinal tract
6. Current communicable disease (e.g. upper respiratory tract infection)
7. Malignant disease and/or patients who are receiving systemic anti-neoplastic agents
8. Psychiatric diseases (e.g. dementia, depression, schizophrenia, autism, Asperger Syndrome) or other incapacity for adequate cooperation
9. Chronic neurological/neurodegenerative diseases (e.g. Parkinson's disease, multiple sclerosis)
10. Autoimmune disease and/or patients receiving immunosuppressive medications
11. Major relevant allergies (e.g. food allergy, multiple allergies)
12. Chronic pain syndromes (e.g. fibromyalgia)
13. Chronic fatigue syndrome
14. Obesity (body mass index>30) or metabolic syndrome
15. Antimicrobial treatment or prophylaxis within the last 3 months
16. Other chronic use of drugs that may affect the microbiome, e.g. proton pump inhibitors
17. Females who are pregnant or breast-feeding
18. Known clinically significant abnormal laboratory values
19. Abuse of alcohol or drugs
20. Probiotic intake within the last 6 weeks
21. Bowel cleansing within the last 6 months
22. Any clinically significant disease/condition which in the investigator's opinion could interfere with the results of the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 10 healthy volunteers will be recruited via local advertisements.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Differences in the composition of the microbiota in luminal and mucosal samples along the large intestine Composition of the microbiota in luminal as well as mucosal samples | 1 day
  16S rRNA-based next generation sequencing

SECONDARY OUTCOMES:
Microbial composition of rectal and faecal microbiota | 1 day
  16S rRNA-based next generation sequencing
Metabolic profile in faecal samples along the intestinal tract | 1 day
  metabolomics
Gene expression of transporters for bacterial products in mucosal biopsies along the colon | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Robert Brummer, Prof., Principal Investigator — Region Örebro County, Örebro University
Locations (1):
- Örebro university, Örebro, Örebro County, Sweden

IPD SHARING:
Plan to Share IPD: No